CLINICAL TRIAL: NCT07321951
Title: A Multicenter, Randomized, Double-blind, Phase II Study to Evaluate the Efficacy and Safety of SHR-1819 Injection in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of SHR-1819 in Patients With Moderate-to-severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1819-207
Record Dates: First submitted 2025-12-21; First posted 2026-01-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1819 Injection Group with Dose 1 (Experimental)
  Interventions: Drug: SHR-1819 Injection; Drug: SHR-1819 Injection Blank Preparation
- SHR-1819 Injection Group with Dose 2 (Experimental)
  Interventions: Drug: SHR-1819 Injection; Drug: SHR-1819 Injection Blank Preparation
- SHR-1819 Injection Group with Dose 3 (Experimental)
  Interventions: Drug: SHR-1819 Injection; Drug: SHR-1819 Injection Blank Preparation

INTERVENTIONS:
Drug: SHR-1819 Injection — SHR-1819 injection.
Drug: SHR-1819 Injection Blank Preparation — SHR-1819 injection blank preparation.

SUMMARY:
This trial was designed to evaluate the efficacy and safety of SHR-1819 in adult patients with moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent, the subjects are ≥18 years old and ≤75 years old, male or female.
2. The subjects have voluntarily signed the informed consent form prior to the start of any procedures related to the study, are able to communicate smoothly with the researcher, understand and are willing to strictly abide by the requirements of this clinical research protocol to complete the study.
3. Topical emollients are applied at a stable dose twice daily for at least 7 days before the first dose in the run-in phase and continued for the duration of the study.
4. Have atopic dermatitis at the time of screening and have an investigator-assessed history of atopic dermatitis for at least 1 year before screening.
5. Have moderate to severe atopic dermatitis during the screening period and on the day of the first dose.

Exclusion Criteria:

1. Have other active skin disease or skin complications due to other conditions that may affect the evaluation of Atopic Dermatitis (AD).
2. A history of spring keratoconjunctivitis and/or atopic keratoconjunctivitis within 6 months prior to screening.
3. Has malignancy or has a history of malignancy.
4. Have serious concomitant diseases and other conditions that the investigator considers inappropriate to participate in this trial.
5. Hypersensitivity to the study drug or any ingredient in the study drug.
6. Females who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who achieved EASI-75 (≥75% decrease in the score on the Eczema Area and Severity Index (EASI) from the baseline). | Week 24.
  Eczema Area and Severity Index score using the Eczema Area and Severity Index scale.

SECONDARY OUTCOMES:
The proportion of participants with a baseline daily Itch Numeric Rating Scale (I-NRS) score of ≤4 per week. | Week 24.
  The Itch Numeric Rating Scale score using the Itch Numeric Rating Scale.
Adverse events (AEs). | About 42 weeks.
The concentration of SHR-1819 in serum. | From week -16 to week -8, about every 4 weeks; From week 0 to week 32, about every 8 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided